CLINICAL TRIAL: NCT02536443
Title: Contemporary Modalities in Treatment of Heart Failure
Acronym: COMMIT-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Mariusz Gasior, Professor, PhD, Silesian Centre for Heart Diseases
Other Study IDs: COMMIT015
Record Dates: First submitted 2015-08-23; First posted 2015-08-31 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure
Keywords: heart failure; prognosis; clinical characteristics
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Contemporary Modalities In Treatment of Heart Failure Registry (COMMIT-HF) is an observational study on an all-comer systolic heart failure population hospitalized in a highly specialized cardiovascular center. The aim of the study is to assess the clinical characteristics, treatment modalities and prognosis in this population.

DETAILED DESCRIPTION:
The Contemporary Modalities In Treatment of Heart Failure Registry (COMMIT-HF) is a single-center observational study that is underway in the 3rd Chair and Department of Cardiology of Silesian Center for Heart Diseases in Zabrze, Poland. Data collection is patient-based (not event-based).

The main objective of the COMMIT-HF Registry is to clarify the overall clinical characteristics of systolic heart failure patients, their demographics and clinical profile, current management, in-hospital outcomes and long-term follow-up, with regard to the administered treatment.

The study population is formed by all-comer patients hospitalized in cardiology wards and intensive cardiac care units with a diagnosis of systolic heart failure. For the purpose of this study heart failure is defined as a set of symptoms resulting from myocardial systolic function impairment, confirmed in resting transthoracic echocardiography with left ventricular ejection fraction (LVEF) ≤35%. Patients with acute coronary syndromes are excluded from the analysis.

Complete patient demographics; medical history, complete hospitalization data (diagnostic and therapeutic) and in-hospital results are collected in an electronic form by the attending physician. The patients are under constant follow-up for all cause mortality and major adverse events.

ELIGIBILITY:
Inclusion Criteria:

* symptom based diagnosis of heart failure
* echocardiographically confirmed impaired left ventricular ejection fraction ≤35%.

Exclusion Criteria:

* acute coronary syndrome on admission
* ≥ 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is formed by all-comer patients hospitalized in cardiology wards and intensive cardiac care units with a diagnosis of systolic heart failure. For the purpose of this study heart failure is defined as a set of symptoms resulting from myocardial systolic function impairment, confirmed in resting transthoracic echocardiography with left ventricular ejection fraction (LVEF) ≤35%.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reported deaths from any cause | From date of inclusion until the date of death from any cause, assessed up to 1 year

SECONDARY OUTCOMES:
Number of participants with reported heart-failure related rehospitalization | From date of inclusion until the date of first event, assessed up to 1 year
Number of participants with reported myocardial infarction | From date of inclusion until the date of first event, assessed up to 1 year
Number of participants with reported cerebrovascular insult | From date of inclusion until the date of first event, assessed up to 1 year
Number of participants to undergo mechanical circulatory support implantation | From date of inclusion until the date implantation, assessed up to 1 year
Number of participants to undergo orthotopic heart transplantation | From date of inclusion until the date transplantation, assessed up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Gasior, Prof., PhD, Principal Investigator — 3rd Chair and Department of Cardiology, Silesian Center for Heart Diseases; Lukasz Pyka, MD, Study Chair — 3rd Chair and Department of Cardiology, Silesian Center for Heart Diseases
Locations (1):
- SIlesian Center for Heart Diseases, Zabrze, Silesian Voivodeship, Poland

REFERENCES:
- [Result] Gasior M, Pyka L, Gorol J, Hawranek M, Tajstra M, Slonka G, Kurek A, Krajewski A, Rozentryt P, Gierlotka M, Lekston A, Zembala M, Polonski L. COnteMporary Modalities In Treatment of Heart Failure: a report from the COMMIT-HF registry. Kardiol Pol. 2016;74(6):523-8. doi: 10.5603/KP.a2015.0224. Epub 2015 Nov 24. PMID 26596896
- [Result] Pyka L, Hawranek M, Tajstra M, Gorol J, Lekston A, Gasior M. Complete percutaneous revascularisation feasibility in ischaemic heart failure is related to improved outcomes: insights from the COMMIT-HF registry. Kardiol Pol. 2017;75(5):453-461. doi: 10.5603/KP.a2017.0018. Epub 2017 Feb 2. PMID 28150287
- [Result] Kurek A, Tajstra M, Gadula-Gacek E, Buchta P, Skrzypek M, Pyka L, Wasiak M, Swietlinska M, Hawranek M, Polonski L, Gasior M, Kosiuk J. Impact of Remote Monitoring on Long-Term Prognosis in Heart Failure Patients in a Real-World Cohort: Results From All-Comers COMMIT-HF Trial. J Cardiovasc Electrophysiol. 2017 Apr;28(4):425-431. doi: 10.1111/jce.13174. Epub 2017 Mar 7. PMID 28176442
- [Result] Wasilewski J, Pyka L, Hawranek M, Tajstra M, Skrzypek M, Wasiak M, Suliga K, Bujak K, Gasior M. Prognostic value of red blood cell distribution width in patients with left ventricular systolic dysfunction: Insights from the COMMIT-HF registry. Cardiol J. 2018;25(3):377-385. doi: 10.5603/CJ.a2017.0037. Epub 2017 Mar 29. PMID 28353308
- [Result] Wasilewski J, Pyka L, Hawranek M, Osadnik T, Kurek A, Skrzypek M, Niedziela J, Desperak P, Kulaczkowska Z, Brzezina M, Krawczyk M, Gasior M. Prognostic value of neutrophil-to-lymphocyte ratio in predicting long-term mortality in patients with ischemic and nonischemic heart failure. Pol Arch Med Wewn. 2016;126(3):166-73. doi: 10.20452/pamw.3316. Epub 2016 Mar 18. PMID 26991886
- [Result] Tajstra M, Pyka L, Gorol J, Pres D, Gierlotka M, Gadula-Gacek E, Kurek A, Wasiak M, Hawranek M, Zembala MO, Lekston A, Polonski L, Bryniarski L, Gasior M. Impact of Chronic Total Occlusion of the Coronary Artery on Long-Term Prognosis in Patients With Ischemic Systolic Heart Failure: Insights From the COMMIT-HF Registry. JACC Cardiovasc Interv. 2016 Sep 12;9(17):1790-7. doi: 10.1016/j.jcin.2016.06.007. PMID 27609252
- [Result] Siedlecki L, Szygula-Jurkiewicz B, Pyka L, Krol B, Szczurek W, Gasior M. Clinical features, management and mortality in diabetic and non-diabetic patients with heart failure - observations from the COMMIT-HF registry. Kardiochir Torakochirurgia Pol. 2017 Sep;14(3):170-174. doi: 10.5114/kitp.2017.70530. Epub 2017 Sep 30. PMID 29181044
- [Result] Szygula-Jurkiewicz B, Siedlecki L, Pyka L, Romuk E, Przybylowski P, Gasior M. Red blood cell distribution width, relative lymphocyte count, and type 2 diabetes predict all-cause mortality in patients with advanced heart failure. Pol Arch Intern Med. 2018 Feb 28;128(2):115-120. doi: 10.20452/pamw.4149. Epub 2017 Nov 9. PMID 29125137